CLINICAL TRIAL: NCT04021745
Title: Mindful Eating - Bringing Awareness Into Eating
Brief Title: Bringing Awareness Into Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1904002405
Record Dates: First submitted 2019-07-15; First posted 2019-07-16 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Stress Eating; Reward-based Eating; Craving-related Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-based mindful eating (Experimental): The intervention will be delivered through a mindful eating smartphone application using the latest evidence-based mindful eating methods and behavior change theory.
  Interventions: Behavioral: App-based mindful eating

INTERVENTIONS:
Behavioral: App-based mindful eating — This is a mindful eating smartphone application comprised of twenty-eight modules of 10-15 minutes each designed to teach mindfulness for binge eating. The feature that is being tested will ask individuals to do a mental exercise when they're craving and will measure their satisfaction related to the experience.

SUMMARY:
The purpose of this study is to test an app-based mindful eating intervention to decrease the reward value of unhealthy food.

DETAILED DESCRIPTION:
Eating healthily is highly beneficial. However, changing eating habits is notoriously difficult. Individuals often believe that they simply need to "restrain" their eating impulses in order to eat more healthily. However, such an approach has not only been shown to be quite ineffective over long time spans, it is also associated with aversive feelings: It simply does not feel good to struggle with one's own impulses.

Investigators are testing a new approach to overcoming unhealthy eating habits, which utilizes mindful eating to change the reward value of unhealthy food. The hypothesis is that if people pay attention to how unhealthy food (e.g. "junk" food) makes them feel in their bodies, their liking it and desire to eat it will decrease naturally. Participants might become aware, for example, that eating a whole bag of chips leads to nausea, while eating a salad makes them feel fresh and energetic.

Investigators will assess whether and how the anticipated and actual satisfaction associated with unhealthy food will decrease the more often participants use this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Craves & overeats a food at least 4 times/week (can be a specific food or food category - i.e. salty or sweet)
2. Desire to change eating habits
3. Owns a smartphone
4. Fluency in English

Exclusion Criteria:

1. Current eating disorder
2. Current strict diet (e.g. paleo, keto, vegan, calorie restriction)
3. Pregnancy
4. Current insulin use
5. Previous use of the EatRightNow application

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Change in Reward Based Eating Drive (RED) Scale | 2 months
  The Reward Based Eating Drive (RED) Scale will be used to assess three dimensions of reward-related eating (lack of satiety, preoccupation with food, and lack of control over eating), in order to comprehensively assess the spectrum of reward-related eating. The RED is a 13-item questionnaire that uses a 5-point Likert scale ranging from 0 ("Strongly Disagree") to 4 ("Strongly Agree"). Scores can range from 0 to 52 and higher scores correspond to higher levels of reward-related eating.

SECONDARY OUTCOMES:
Change in Salzburg Stress Eating Scale (SSES) | 2 months
  The Salzburg Stress Eating Scale (SSES) will be used to assess stress eating. The SSES is a 10-item questionnaire that uses a 5-point Likert scale where 1 is "I eat much less than usual" and 5 is "I eat much more than usual". Scores can range from 10 to 50 and higher scores correspond to higher levels of stress eating.
Change in Food Craving Questionnaire - Trait, Reduced (FCQ-T-r) | 2 months
  Food Craving Questionnaire will be used to assess food cravings. The The FCQ-T-r is a 15-item questionnaire that uses a 5-point Likert scale where 1 is "Strongly Disagree" and 5 is "Strongly Agree". Scores can range from 15 to 75 and higher scores correspond to higher levels of food craving.

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No